CLINICAL TRIAL: NCT07331896
Title: Examining Strategy Training for Optimizing Awareness in Rehabilitation for Community-dwelling Individuals With Spatial Neglect
Brief Title: Strategy Training for Optimizing Awareness in Rehabilitation for Individuals With Spatial Neglect Living
Acronym: SOAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Emily Grattan, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY25090119
Record Dates: First submitted 2025-12-26; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Neglect, Hemispatial
MeSH Terms: conditions — Stroke; Perceptual Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy Training (Experimental): The strategy training intervention teaches individuals to develop personalized goals, self-assess their performance of daily activities, and develop and evaluate strategies designed to overcome barriers and improve their performance of daily activities. Participants use a workbook to support their application of the strategy training.
  Interventions: Behavioral: Strategy Training
- Attention Control (Active Comparator): The attention control intervention controls for the non-specific effects of strategy training. The study team will administer the standardized and dose-matched protocol, using scripted open-ended questions to facilitate participants' reflections on their rehabilitation activities and experiences. Participants complete a daily journal, merely reviewing their rehabilitation activities.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Strategy Training — This intervention will use an adapted form of strategy training for people with neglect.
  Arms: Strategy Training
Behavioral: Attention Control — This intervention will use a reflective listening protocol.
  Arms: Attention Control

SUMMARY:
It is common for individuals after stroke to have a cognitive perceptual impairment called unilateral spatial neglect (neglect). Individuals with neglect have difficulty paying attention to one side of their body or one side of the environment and therefore experience difficulty performing daily activities. There are a lack of effective treatments for neglect and new interventions are needed to help reduce disability for these individuals. Metacognitive strategy training (strategy training) is an intervention that has the potential to reduce neglect-related disability and improve individuals' awareness of their neglect. This study seeks to examine the effects of strategy training on self-awareness, disability, and neglect specifically for individuals who are living in the community after their stroke.

DETAILED DESCRIPTION:
Unilateral spatial neglect (neglect) post stroke is characterized by a lack of attention to one side of the body or one side of the environment. Individuals with neglect experience significant disability and are often unaware of their neglect symptoms which can make it even more difficult to treat. There are a lack of effective treatments for neglect and new interventions are needed to help reduce disability for these individuals. Metacognitive strategy training (strategy training) is an intervention that has the potential to reduce neglect-related disability and improve individuals' awareness of their neglect. Strategy training teaches individuals to develop personalized goals, self-assess their performance of daily activities, and develop and evaluate strategies designed to overcome barriers and improve their performance of daily activities. While strategy training shows promise for individuals with neglect, no studies have tailored the intervention for this group of individuals or examined the effects of strategy training for individuals with neglect specifically with individuals living in the community. This study examines whether strategy training facilitates reductions in disability and neglect and improves self-awareness after stroke.

ELIGIBILITY:
Inclusion Criteria:

* had a stroke
* presence of neglect as determined by score of <18 or 2 or more collisions on the Virtual Reality Lateralized Attention Test (VRLAT) or score below established cutoff for neglect on one of the six subtests of the Behavioral Inattention Test (BIT);
* score of 4 or higher on any item of the Self-Regulation Skills Interview (SRSI)
* ≥18 years old
* lives within 30 miles of the University of Pittsburgh in a community dwelling.

Exclusion Criteria:

* Boston Diagnostic Aphasia Examination (BDAE) Severity Scale score of 0
* dementia per medical record
* active major depressive disorder per medical record
* not willing to be videotaped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in self-awareness | Baseline to Post-intervention (up to 4 weeks)
  Change in self-awareness measured with the Catherine Bergego Scale. The Catherine Bergego Scale includes a therapist-rated assessment and client-rated (self) assessment. Total scores on the Catherine Bergego Scale therapist-rated assessment and client-rated (self) assessment each range from 0-30 (higher=greater neglect). The difference in client-rated total Catherine Bergego Scale scores and assessor-rated total Catherine Bergego Scale scores will be used as a measure of self-awareness (smaller difference=better awareness). The a priori criterion for change was a medium effect size of change (Cohen's d≥0.5)

SECONDARY OUTCOMES:
Client Satisfaction with Strategy Training | Post-intervention (up to 4 weeks)
  Client satisfaction is measured using the Client Satisfaction Questionniare-8. The a priori criterion for satisfaction was: ≥90% of participants report mean satisfaction score ≥3 on the Client Satisfaction Questionnaire-8 items. Item scores on the Client Satisfaction Questionnaire-8 range from 0-4. Higher scores on the Client Satisfaction Questionnaire-8=greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Grattan, PhD, OTR/L, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
At present, there is no plan to share data.